CLINICAL TRIAL: NCT05980377
Title: Patterns of Hemophilia Care in Patients Admitted in Assiut Children University Hospital
Brief Title: Patterns of Hemophilia Care in Assiut Children Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Ahmed Abd El-Bary, Principal Investigator, Assiut University
Other Study IDs: Pattern of Hemophilia care
Record Dates: First submitted 2023-07-29; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Hemophilia A; Hemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

SUMMARY:
Hemophilia A and B are congenital, recessive X-linked disorders caused by lack or deficiency of clotting factor VIII (FVIII) or IX (FIX), respectively. The severity of the disease depends on the reduction of levels of FVIII or FIX, which are determined by the type of the causative mutation in the genes encoding the factors (F8 and F9, respectively). The hallmark clinical characteristic, especially in untreated severe forms, is bleeding (spontaneous or after trauma) into major joints such as ankles, knees and elbows, which can result in the development of arthropathy. Intracranial bleeds and bleeds into internal organs may be life-threatening. The median life expectancy was ~30 years until the 1960s, but improved understanding of the disorder and development of efficacious therapy based on prophylactic replacement of the missing factor has caused a paradigm shift, and today individuals with hemophilia can look forward to a virtually normal life expectancy and quality of life.

DETAILED DESCRIPTION:
Hemophilia A and B are congenital, recessive X-linked disorders caused by lack or deficiency of clotting factor VIII (FVIII) or IX (FIX), respectively. The severity of the disease depends on the reduction of levels of FVIII or FIX, which are determined by the type of the causative mutation in the genes encoding the factors (F8 and F9, respectively). The hallmark clinical characteristic, especially in untreated severe forms, is bleeding (spontaneous or after trauma) into major joints such as ankles, knees and elbows, which can result in the development of arthropathy. Intracranial bleeds and bleeds into internal organs may be life-threatening. The median life expectancy was ~30 years until the 1960s, but improved understanding of the disorder and development of efficacious therapy based on prophylactic replacement of the missing factor has caused a paradigm shift, and today individuals with hemophilia can look forward to a virtually normal life expectancy and quality of life.

Historically, hemophilia treatment has focused on replacement of the missing coagulation factor to achieve hemostasis. Treatment progressed from use of cryoprecipitate (FVIII replacement in HA) or fresh frozen plasma (FFP) to plasma-derived factor concentrates, allowing for early control of hemorrhage, home therapy and accessibility for the introduction of prophylaxis. Contamination of factor concentrate supply with human immunodeficiency virus and hepatitis C virus led to the unfortunate infection of most of the severe hemophilia population in the 1980s, necessitating development of improved methods to screen and inactivate viruses. These mechanisms include dry-heat, pasteurisation, solvent-detergent treatment, immunoaffinity purification and nanofiltration, although some risk from emerging infections remains. Recombinant factor therapies were introduced to address the concern for infection transmission but raised new challenges regarding the risk of inhibitor formation. The extended half-life (EHL) factor products are a result of engineering proteins for longer recovery times in persons with hemophilia (PwH), to reduce frequency of dosing for prophylax

-Factor VIII mimetic Emicizumab (Hemlibra, Genentech/Roche) is a first in-class humanised bispecific antibody substitution for HA designed to function as FVIIIa by binding one arm of the antibody to FIXa and the other arm to FX, accelerating activation of Fxa and propagating thrombin production. The application and incorporation of this novel approach using a SC antibody to prevent bleeding was outlined in a series of clinical trials (HAVEN) including PwHA with inhibitors, paediatric PwHA with inhibitors and PwHA without inhibitors. The bispecific antibody mechanism and half-life (˜28 days) overcomes the inhibitory alloantibody, limits the need for IV access and decreases infusion frequency. In HAVEN-1, males with severe HA and inhibitors aged ≥12 years received weekly prophylaxis (1·5 mg/kg) with emicizumab and had an 87% reduction in overall annualized bleeding rate (ABR)

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with hemophilia attending Assiut university hospital of children

Exclusion Criteria:

* Any patient with other bleeding disorder

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All patients diagnosed with hemophilia attending Assiut university hospital of children in 2 years duration
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
care in hemophilia patients | Baseline
  Describe different aspects of care in hemophilia patients in Assiut children university hospital
Describe complications in availability of factors | Baseline
  describe different aspects of complications and challenges in availability of factors ,bypassing agents which are used to manage hemophilia patients with inhibitors in Assiut children university hospital